CLINICAL TRIAL: NCT05218317
Title: Evaluation of Relapse Presence in Multiple Sclerosis Patients by Cross-Sectional In-Vivo Corneal Confocal Microscopy
Brief Title: Evaluation of Relapse Presence in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.240
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis Relapse
Keywords: multiple sclerosis, in-vivo corneal confocal microscopy, relapse, inflammation, neurodegeneration, neuroregeneration
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Recurrence; Inflammation; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MS-Relapse: Twenty-seven patients (MS-Relapse) for whom the administration of intravenous corticosteroids was decided due to the diagnosis of new relapse.
  The diagnosis of RRMS and the new relapse was confirmed and decided by a senior neurologist (K.A) of Marmara University Department of Neurology, according to the revised McDonald criteria, based on clinical and radiological findings These subjects underwent Corneal Confocal Microscopy (IVCM).
  Interventions: Diagnostic Test: in-vivo Corneal Confocal Microscopy
- MS-Control: Thirty-one patients (MS-Control) who were followed up with the diagnosis of RRMS The diagnosis of RRMS and the new relapse was confirmed and decided by a senior neurologist (K.A) of Marmara University Department of Neurology, according to the revised McDonald criteria, based on clinical and radiological findings.
  These subjects underwent Corneal Confocal Microscopy (IVCM).
  Interventions: Diagnostic Test: in-vivo Corneal Confocal Microscopy
- Healthy Controls: Thirty healthy age and gender similar population These subjects underwent Corneal Confocal Microscopy (IVCM).
  Interventions: Diagnostic Test: in-vivo Corneal Confocal Microscopy

INTERVENTIONS:
Diagnostic Test: in-vivo Corneal Confocal Microscopy — All study subjects underwent IVCM (Rostock Cornea Module, Heidelberg Retinal Tomograph III; Heidelberg Engineering, Germany). Before the examination, two drops of topical anesthetic with proparacaine hydrochloride (Alcaine 0.5%, Alcon-Couvreur, Belgium) were applied to both eyes. A carbomer-based gel (Viscotears 0.2%; Dr. Gerhard Mann, Chem.- Pharm. Fabrik, Germany) was used as the coupling agent between the cornea and the applanating cap of IVCM. For correctly positioning the central cornea, all subjects were asked to fixate a determined fixation point and controlled with the device camera. All scans were performed in approximately 5 minutes for each eye by a single experienced ophthalmologist, masked from the subject's disease status.

SUMMARY:
Purpose: This study aims to investigate the demonstrability of increased inflammation and neurodegeneration in multiple sclerosis (MS) patients in relapse period compared to MS patients in remission by cross-sectional analysis of in-vivo corneal confocal microscopy (IVCM), and to evaluate the alternations with a second IVCM administered at least 6 months after the relapse period.

Methods: This prospective, non-randomized-controlled, cross-sectional study included 58 MS patients which were grouped regarding the presence of relapse (MS-Relapse group [n=27] and MS-Control group [n=31]), and age-sex matched 30 healthy controls (HC). The corneal nerve fiber density (CNFD), the corneal nerve branch density (CNBD), the corneal nerve fiber length (CNFL), and dendritic cell (DC) density were evaluated in all MS patients and HCs by IVCM. If the patients in the MS-relapse group did not have an attack within 6 months, the same parameters were evaluated with the second IVCM. The patients with a history of optic neuritis or trigeminal symptoms were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom the administration of intravenous corticosteroids was decided due to the diagnosis of new relapse
* Patients who were followed up with the diagnosis of RRMS
* Healthy controls

Exclusion Criteria:

* Being younger than 18 years old
* Having any other neurological or metabolic diseases
* Ophthalmological diseases
* A history of optic neuritis and trigeminal symptoms
* Ocular trauma or surgery
* Contact lens use
* The patients who had a relapse attack 6 months prior to the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty-eight patients with RRMS and 30 HCs were included in the study. The RRMS patients were divided into two subgroups: 1) Thirty-one patients (MS-Control) who were followed up with the diagnosis of RRMS, 2) Twenty-seven patients (MS-Relapse) for whom the administration of intravenous corticosteroids was decided due to the diagnosis of new relapse.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Corneal nerve fiber density (CNFD) | Baseline
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFD.
Corneal nerve fiber density (CNFD) | 6 Month
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFD.
Corneal nerve branch density (CNBD) | Baseline
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNBD.
Corneal nerve branch density (CNBD) | 6 Month
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNBD.
Corneal nerve fiber length (CNFL) | Baseline
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFL.
Corneal nerve fiber length (CNFL) | 6 Months
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFL.

SECONDARY OUTCOMES:
Dendritic Cells | Baseline
  the number of DCs counted by ImageJ's Cell Counter plug-in
Dendritic Cells | 6 Months
  the number of DCs counted by ImageJ's Cell Counter plug-in

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)